CLINICAL TRIAL: NCT06403514
Title: An Experimental Examination of a Racecar-simulation Psychoeducational Intervention and the Effects on Health and Performance-based Outcomes of Veterans Diagnosed With PTSD
Brief Title: The Effects of a Psychoeducational Intervention on Health and Performance-based Outcomes of Veterans Diagnosed With PTSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Southeastern University (Other)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Principal Investigator, William Edmonds, Professor, Nova Southeastern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-210-NSU
Record Dates: First submitted 2024-04-22; First posted 2024-05-08 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Post Traumatic Stress Disorder
Keywords: Veterans
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: The design is a single-case approach with the application of range-bound changing criterion design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Trial (Experimental): Psychological Skills Training (PST). The PST will include elements, both generalized and idiosyncratic, for each participant and is considered an adapted model of stress inoculation skills training protocol. The specifics will include each participant's unique optimal and poor ranges of performance (i.e., IZOFs), which will be calculated utilizing HRV, BPM, EMG, respiration and subjective affect. The participants will be introduced to their IZOFs and then taught general and specific approaches to self-regulation using elements of a mindfulness protocol for BFB in a clinical environment. A dual-monitor setup for the BFB application will be employed.
  Interventions: Other: Psychological Skills Training (PST)

INTERVENTIONS:
Other: Psychological Skills Training (PST) — PST will include self-talk, imagery, goal-setting and arousal regulation (Biofeedback)

SUMMARY:
Nova Southeastern University and the Veterans trust through this line of research will strengthen community engagement and awareness for the need to recognize and provide treatment models for veterans diagnosed with PTSD. The goal is to improve self-regulatory mechanisms within the racecar simulated-environment with the hope it translates to real-life scenarios.

The design is a single-case approach with the application of range-bound changing criterion design. It will include elements of stress-inoculation therapy, cognitive processing therapy, optimal zones of functioning, biofeedback and psychological skills training. This particular design will allow for the collection and identification of the idiosyncratic differences between each participant which will guide how the data are collected and the tailoring of the intervention.

DETAILED DESCRIPTION:
Initially, the participants undergo all pre-test assessments at the Neuropsychology Assessment Center prior to being deemed eligible for the experiment. Next, participants will be scheduled individually to visit the Race Lab to become acquainted with the lab and virtual environment. Basics of the research study will be explained to each participant as part of the adaptation process. This will include a brief educational lesson on the Psychological Skills Training intervention. Following the adaptation period, the participant will commence with the experimental race-car psychoeducational intervention.

Design. A single-case approach with the Range-Bound Changing Criterion design (RBCC) will used. The RBCC design is a variant of the changing criterion design used in single-subjects research to allow for the systematic shaping of behaviors in the pursuit of short- and long-term based objectives. As a result, the design adequately allows for the application of the Learning-Modification-Application Model (LMA), which is based on the premise of periodization (i.e., step-wise incremental changes as a means to improve performance through increased challenges). That is, following baseline collection, a performance range-bound criterion will be established a-priori based on the phase of the LMA model. Control is established when the participant's performance consistently matches or surpasses the criterion within the given phase of the LMA and continues to progress throughout the subsequent intervention phases as performance criteria becomes more rigorous. See Table 1 and Figure 1 for the basics of the RBCC Design.

Table 1. Range-Bound Changing Criterion Design Legend Design Notation Design Phase A Baseline B Learning C Modification D Application

Figure 1. Condensed Design Structure of the RBCC Design

Treatment Phase Design Structure

Learning: A-B-A-B-A-B-A-B-A-B-A

Modification: A-C-A-C-A-C-A-C-A-C-A

Application: A-D-A-D-A-D-A-D-A-D-A

Procedural Steps. There are three main phases of the experiment- Learning, Modification and Application. Within the Learning and Modification phases, participants will be required to complete five separate time-trials (i.e., race against the clock in the absence of other competitors), with each trial consisting of four laps. Multiple checkpoints within the race along with the finish line will allow performance times to be collected. The Application phase will also include five separate time trials, but the race will include competitors.

Throughout the experiment, the participant will be connected to physiological recording devices and data will be collected via the baseline and in-trial activities, which include heart rhythms (Beats per minute (BPM) and Heart Rate Variability - (HRV)), Electromyograph (EMG), respiration, and subjective perceptions of affect. Following each experimental phase, immersion, cognitive and somatic anxiety measures will be taken along with self-efficacy. Objective and subjective data from the trials will be reduced and Individual Zone of Optimal Functioning (IZOFs) will be determined to be utilized in the Psychological Skills Training aspect of the experiment.

Psychological Skills Training (PST). The primary focus of PST is to assist the participants in acquiring adequate self-regulatory and coping skills as a mean to increase the participants' coping repertoire.

ELIGIBILITY:
Inclusion Criteria:

* All veterans of the US Military
* Clinical diagnosis of PTSD
* Completed the Veterans Trust Self-Regulatory Mastery course with the Race-Simulator

Exclusion Criteria:

* Severe/markedly elevated severity rating on the CAPS-5
* Extreme/incapacitating severity rating on the CAPS-5
* Asthma
* Emphysema
* Chronic obstructive pulmonary disease
* History of heart disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2024-08-16 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-08-26 (Actual)

PRIMARY OUTCOMES:
The Quality of Life Scale | pre-intervention, immediately after the intervention
  (QOLS). The QOLS is used to assess quality of life across a wide-range of clinical and non-clinical groups and is considered distinct from health status or other indicators of quality of life. Scores range from 16 to 112. Higher scores represent enhanced QOL.
The Difficulties in Emotion Regulation Scale | pre-intervention, immediately after the intervention
  (DERS). The DERS is an assessment tool for gauging challenges in emotion regulation. It allows for the assessment of respondents' interactions with their emotions and generates scores across six distinct subscales. Scores range from 36 to 180. Higher scores represent enhanced self-regulatory skills.
Emotional Self-Efficacy | pre-intervention, immediately after the intervention
  (ESE). ESE is designed to assess an individual's belief that he or she can appropriately respond to positive and negative environmental cues, particularly when there is little motivation to do so. Scores range from 10 to 50. Higher scores represent enhanced emotional efficacy.
The General Self-Efficacy Scale | pre-intervention, immediately after the intervention
  (GSE). The GDE is a 23-item tool based on Bandura's social cognitive theory, measuring overall confidence in life activities with subscales for general (GSE) and social (SSE) self-efficacy. Higher scores predict success in various areas (e.g., vocational, educational, and military settings). Scores range from 10 to 40. Higher scores represent enhanced general efficacy.
Psychological Skills Training Self-Efficacy | pre-intervention, immediately after the intervention
  (PST-SE). Each item of the Psychological Skills Training program will be represented in the PST-SE which include: Arousal Regulation, Self-Talk, Imagery, Goal Setting and Imagery. Scores range from 10 to 40. Higher scores represents enhanced PST efficacy.
The Clinician-Administered PTSD Scale | pre-intervention, immediately after the intervention
  (CAPS-5). The CAPS-5 is a diagnostic interview for assessing post-traumatic stress disorder (PTSD). CAPS is a criterion measure, and it evaluates all PTSD criteria and associated features like dissociation. The results from the CAPS provides global ratings for distress, impairment, response validity, symptom severity, and improvement since the last assessment.
  0. Absent:
  1. Mild / subthreshold:
  2. Moderate / threshold:
  3. Severe / markedly elevated:
  4. Extreme / incapacitating:
  Lower score represents lowered PTSD symptoms.
The Trauma Symptoms Inventory-2-A | pre-intervention, immediately after the intervention
  (TSI-2). The TSI-2 is a self-report tool with 126 items assessing post-traumatic stress and psychological outcomes from traumatic events in adults. The tool is used to assess PTSD symptoms and broader psychological effects (i.e., well-being). Scores range from 0 to 378. Lower scores represent lowered trauma symptoms.

SECONDARY OUTCOMES:
The affect grid | pre-intervention, immediately after the intervention
  (AG). The affect grid is a 9-by-9 grid designed to measure dimensions of perceived physiological arousal and pleasure. The vertical dimension represents arousal and ranges and the horizontal dimension represents pleasure and ranges. Pleasure ranges from 1-9 and Arousal ranges from 1-9. Scores are not qualified as good or bad.
The Immersive Tendency Questionnaire | immediately after the intervention
  (ITQ). The ITQ is designed to assess the subjective experience of being in one place or environment, particularly in a virtual environment. Scores range from 32 to 224. Higher scores represent enhanced perceptions of immersion.

OTHER OUTCOMES:
Performance | pre-intervention, immediately after the intervention
  Performance will be assessed by measuring the time it takes to complete the race trial through each checkpoint. Each phase will consist of five trials and each trial will be comprised of multiple checkpoints including the finish line, which provides recorded performance times. Performance is measures in minutes and seconds it takes to complete each round. Lower performance represents improvements.

CONTACTS AND LOCATIONS:
Overall Officials: William A Edmonds, PhD, Principal Investigator — Nova Southeastern University
Locations (1):
- Nova Southeastern University, Davie, Florida, United States